CLINICAL TRIAL: NCT01150721
Title: Comparing Expectorated and Induced Sputum and Pharyngeal Swabs for Cultures, AFB Smears, and Cytokines in Pulmonary Nontuberculous Mycobacterial Infection
Status: Completed | Type: Observational
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Responsible Party: Sponsor
Other Study IDs: 100149; 10-CC-0149
Record Dates: First submitted 2010-06-24; First posted 2010-06-25 (Estimated); Last update posted 2026-02-05 (Actual); Status verified 2026-02-02

CONDITIONS: Mycobacterium Infections, Non-tuberculous
Keywords: Computerized Tomography; Colony Forming Units; Cystic Fibrosis; Analysis of Variance; Forced Expiratory Volume; Natural History
MeSH Terms: conditions — Mycobacterium Infections; Cystic Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 1/PNMI: Adult patients with Pulmonary Nontuberculous Mycobacterial Infection
- 2/Healthy Volunteers: Healthy Volunteer adults

SUMMARY:
Background:

- Pulmonary nontuberculous mycobacterial infection is a respiratory infection that is sometimes difficult to diagnose. Proper diagnosis depends on accurate collection of respiratory secretions, but these secretions may be contaminated by bacteria present in the mouth at the time of collection. In addition, some individuals may have difficulty providing respiratory secretions, because the infection affects lung function and sputum production. By collecting new samples from individuals who have already been diagnosed with this infection, and comparing the methods of collection, researchers hope to better understand and improve the ability to accurately diagnose and treat the infection at an early stage.

Objectives:

- To compare throat cultures and coughed-up and induced phlegm or sputum in individuals with pulmonary nontuberculous mycobacterial infection and inflammation.

Eligibility:

- Individuals between 18 and 79 years of age who have been diagnosed with pulmonary nontuberculous mycobacterial infection and are currently participating in selected NIH protocols on this infection.

Design:

* The study will require a single 90-minute visit to provide research specimens.
* Participants must not eat or drink for 2 hours prior to the collection of the early morning respiratory specimens. Blood pressure, temperature, pulse, breathing rate, and oxygen saturation level readings will be taken on the day of collection to ensure that participants may safely provide the specimens.
* Participants will provide the following samples:
* Blood sample: Participants will provide a blood sample to measure indicators of inflammation in the blood.
* Throat swab: Participants will brush their teeth thoroughly before allowing researchers to swab the inside of their throat with a sterile swab.
* Sputum collection (regular and induced): Participants will brush their teeth thoroughly and then provide both a regular sputum sample (produced normally) and an induced sputum sample (produced after using a nebulizer to stimulate sputum production).
* No treatment will be provided as part of this protocol.

DETAILED DESCRIPTION:
In this protocol, a repeated measure design is used to examine microbial and molecular results in subjects with a diagnosis of pulmonary nontuberculous mycobacterial infection. Patients often experience difficulties in the spontaneous expectoration of sputum free from contamination with oral flora which contributes to the poor quality of some respiratory specimens sent to the laboratory. At present, it is not known how induced sputum, expectorated sputum, and pharyngeal swabs compare for acid fast bacilli (AFB) smear and culture results. Appropriate specimens are needed in the clinical setting for optimum diagnosis. In this study, procedures for the non-invasive collection of respiratory secretions will be used to decrease risk of specimen contamination.

Subjects who cannot produce respiratory secretions will be compared to patients who are successful. It is not known which factors prevent production of respiratory secretions for testing. Airway inflammation may contribute to difficulty in producing sputum along with dyspnea, phase of illness (newly diagnosed or chronic infection), treatment status, and respiratory condition severity.

Subjects will be characterized by phase of illness determined by health history and inflammation using common laboratory tests of inflammation. Respiratory specimens and blood will be collected for microbial testing and a portion will be stored then tested for analysis of pro-inflammatory cytokines (IL-1, IL-6, IL-8, TNF-alpha, & IFN-gamma). Clinical, demographic, laboratory, and patient subjective variables will be tested using regression statistical methods to determine predictors for specimen production success. Clinical variables to be tested include forced expiratory volume at one minute (FEV1) from a pulmonary function test (PFT), phase of illness and treatment, and age. The laboratory tests indicating inflammation include erythrocyte sedimentation rate (ESR), C-reactive protein (CRP), and Beta-2-Microglobulin (Beta-2M). Patient assessments for dyspnea will be evaluated using the Borg questionnaire.

ELIGIBILITY:
* INCLUSION CRITERIA:

Subjects with PNTM must meet the following criteria to participate in this study:

1. Ages 18-99 years
2. Diagnosis of PNTM
3. Participating on an existing NIH protocol.
4. Willing to allow the proposed protocol to use test results from the protocols. These data include: AFB smear and NTM cultures, HIV testing by ELISA and Western blot testing, CRP, ESR, & Beta-2M, FEV1, and Borg Questionnaire results (Appendices E).

Healthy volunteers must meet the following criteria to participate in this study:

1. Ages 18-80 years
2. Healthy
3. Willing to have blood tests for CRP, Beta-2 M, ESR, and cytokine assessments in respiratory secretions and blood
4. Willing to donate respiratory secretions and blood to be used for future research

EXCLUSION CRITERIA:

Subjects with PNTM:

1. Inability or unwillingness to provide any specimens: blood or respiratory (subjects able to provide blood and at least one type of respiratory secretions will not be withdrawn from the study)
2. Current medications of colony stimulating factors, IFN-gamma, IFN-alpha or monoclonal antibodies such as Rituximab within three months of this study
3. Vital signs falling beyond the following parameters prior to specimen collection procedures:

   1. Temperature (tympanic) greater than 101 degrees Fahrenheit (38.3 degrees Celsius) pulse less than 51 per minute or greater than 124 per minute
   2. Respiratory rate less than 12 per minute or greater than 40 per minute.
   3. Oxygen saturation less than 92 percent
4. New (less than or equal to 30 days) tracheostomy tube, chest tube, or major surgery.
5. Current infection with TB or HIV:

   * Any condition in the judgment of the investigators that would place subjects at risk or would jeopardize the study.

HEALTHY VOLUNTEER PARTICIPANT EXCLUSION CRITERIA:

1. Inability or unwillingness to provide any specimens: blood or respiratory (subjects able to provide blood and at least one type of respiratory secretions will not be withdrawn from the study)
2. Current use of specific biological medications: colony stimulating factors, IFN- >=, IFN- or monoclonal antibodies such as Rituximab within three months of this study
3. Vital signs falling beyond the following parameters prior to specimen collection procedures:

   1. Temperature (tympanic) greater than 101degrees Fahrenheit (38.3 o Celsius)
   2. Pulse less than 51 per minute or greater than 124 per minute
   3. Respiratory rate less than 12 per minute or greater than 40 per minute.
   4. Oxygen saturation less than 92%
4. Recent (less than or equal to 30 days) tracheostomy tube, chest tube, or major surgery.
5. Current infection with tuberculosis
6. History of chronic lung disease associated with increased inflammation to include: asthma, chronic obstructive pulmonary disease, pulmonary fibrosis, or any lung condition that, in the opinion of the investigator, may potentially be associated with an increased pulmonary inflammatory response.
7. Any condition in the judgment of the investigators that would place subjects at risk or would jeopardize the study.

   Participation of Women:

   Contraception:

   -The protocol has no requirement for contraception or restriction due to contraception choice as the study interventions (blood draw and collection of respiratory secretions have no restriction relative to contraception).

   Pregnancy:

   -The protocol has no requirement for restriction due to pregnancy. Study interventions (blood draw and collection of respiratory secretions have no restrictions relative to pregnancy.

   Participation of Minorities:

   -There are no restrictions for minority participation in this study.

   Participation of Children:

   -Children are not included in this study since the benefit versus the procedural burden of the protocol does not support their inclusion. Asking children to produce three respiratory specimens at a protocol visit is thought to be burdensome. Infants and young children cannot spontaneously expectorate. The main protocol upon which this protocol recruits only includes adults.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Healthy adult volunteers and adult patients with Nontuberculous Mycobacterial Infection
Sampling Method: Non-Probability Sample
Enrollment: 177 (Actual)
Dates: Start 2010-11-10 (Actual)

PRIMARY OUTCOMES:
Compare collection methods in respiratory secretions | Day 1
  Compare three standardized non-invasive collection methods for obtaining respiratory secretions

SECONDARY OUTCOMES:
Characterize subjects by phase of illness, status of medications and inflammation | Day 1
  Common blood laboratory tests of inflammation
Compare molecular markers of inflammation | Day 1
  Expectorated and induced sputum, pharyngeal swabs, and blood in order to characterize inflammation in two groups of participants with PNTM: 1. patients currently culture positive for NTM infection, 2. patients currently NTM culture negative and in healthy volunteers
Determine predictors for success with production of respiratory secretions | Day 1
  Expectorated and induced sputum

CONTACTS AND LOCATIONS:
Overall Officials: Steven M Holland, M.D., Principal Investigator — National Institutes of Health Clinical Center (CC)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2010-CC-0149.html